CLINICAL TRIAL: NCT07140250
Title: Shared Decision-Making With ChatGPT for Patients With Sinusitis and Nasal Obstruction
Brief Title: Using ChatGPT to Help Guide Treatment for Sinus and Nasal Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carol Yan (Other)
Responsible Party: Sponsor-Investigator, Carol Yan, Associate Professor of Otolaryngology, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 810119
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Sinusitis; Nasal Obstruction; Rhinitis
Keywords: sinusitis; shared decision making; rhinitis; chatGPT; nasal obstruction
MeSH Terms: conditions — Sinusitis; Nasal Obstruction; Rhinitis | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared Decision Making on Sinusitis Treatment Facilitated by ChatGPT (Active Comparator): Shared decision making (SDM) about sinusitis treatment will be facilitated by ChatGPT through participant driven question and answers using AI support via ChatGPT
  Interventions: Other: Education with AI Technology
- Shared Decision Making on Sinusitis Treatment Facilitated by Google (Placebo Comparator): Shared decision making (SDM) about sinusitis treatment will be facilitated by traditional internet search engines (Google) with AI mode off. Participate education on sinusitis treatment will be driven by traditional internet searches
  Interventions: Other: Education using Traditional Internet Search Engines

INTERVENTIONS:
Other: Education with AI Technology — Shared decision making (SDM) about sinusitis treatment will be facilitated by AI technology via ChatGPT
  Arms: Shared Decision Making on Sinusitis Treatment Facilitated by ChatGPT
Other: Education using Traditional Internet Search Engines — Participant Education in Sinusitis using Traditional Internet Search Engines through Google
  Arms: Shared Decision Making on Sinusitis Treatment Facilitated by Google

SUMMARY:
The goal of this clinical trial is to evaluate whether ChatGPT can improve shared decision-making by increasing treatment-related knowledge and reducing decisional conflict in adult patients with chronic rhinosinusitis (CRS) or nasal obstruction who have been deemed candidates for surgery.

The main questions it aims to answer are:

* Does ChatGPT improve patient understanding of CRS/nasal obstruction treatment options compared to widely utilized web searches?
* Does ChatGPT reduce decisional conflict regarding surgical versus medical management compared to traditional search engine? Researchers will compare a group using Google (standard internet search with AI turned off) after standard counseling to a group using ChatGPT after standard counseling to see if ChatGPT leads to higher knowledge scores, lower decisional conflict scores, and higher satisfaction with the information platform.

Participants will:

* Complete baseline surveys assessing demographics, treatment-related knowledge, and decisional conflict
* Be randomized to use either Google or ChatGPT to research their surgery for 10 minutes after standard in-office counseling
* Complete follow-up surveys assessing knowledge, decisional conflict, and satisfaction with the information source
* Allow the research team to review their medical record for relevant clinical history and disease-specific quality-of-life scores (SNOT-22)

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or older) UC San Diego Health System Rhinology patients
* Diagnosis of chronic rhinosinusitis and/or nasal obstruction based on clinical criteria or radiologic evidence
* Planning to pursue surgical intervention for CRS or nasal obstruction
* Ability to complete online survey in English or Spanish

Exclusion Criteria:

* Unable to complete survey assessments online via REDCap
* Under the age of 18 years
* Vulnerable patient populations such as those who are pregnant and institutionalized individuals
* Patients with benign and malignant tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Decisional Conflict Scale (DCS) score | Immediate - Following completion of education using AI vs traditional education
  Change in Decisional Conflict Scale (DCS) score

SECONDARY OUTCOMES:
System usability scale (SUS) scores | Immediate following education
Score on treatment-related knowledge questionnaire (MCQ) | Immediate following education

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided